CLINICAL TRIAL: NCT04810130
Title: Effect of Repetitive Soccer Heading on Biomechanics and Physiological Measures
Brief Title: Physiological Effects of Soccer Heading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-017267
Record Dates: First submitted 2021-03-04; First posted 2021-03-22 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Repeated Head Impacts
Keywords: Soccer Heading

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kicking (Sham Comparator): Subjects will complete a suite of clinical and neurophysiological assessments at 3 timepoints (Pre, 0-hour post, and 16-72 hour post soccer kicking intervention).
  Interventions: Other: Soccer Kicking
- Soccer Heading (Frontal) (Experimental): Subjects will complete a suite of clinical and neurophysiological assessments at 3 timepoints (Pre, 0-hour post, and 16-72 hour post soccer heading intervention).
  Interventions: Other: Soccer Heading (Frontal)
- Soccer Heading (Oblique) (Experimental): Subjects will complete a suite of clinical and neurophysiological assessments at 3 timepoints (Pre, 0-hour post, and 16-72 hour post soccer heading intervention).
  Interventions: Other: Soccer Heading (Oblique)

INTERVENTIONS:
Other: Soccer Kicking — Subjects assigned to the soccer kicking arm will complete 10 soccer kicks in 10 minutes.
  Arms: Kicking
Other: Soccer Heading (Frontal) — Subjects assigned to the soccer heading (frontal) arm will complete 10 frontal soccer headers (ball headed directly back to launch direction) in 10 minutes. Soccer balls will be projected at 10-17.5 m/s from approximately 10-15 m with a JUGS ball launcher.
  Arms: Soccer Heading (Frontal)
Other: Soccer Heading (Oblique) — Subjects assigned to the soccer heading (oblique) arm will complete 10 oblique soccer headers (ball headed 90° to the right from ball launch direction) in 10 minutes. Soccer balls will be projected at 10-17.5 m/s from approximately 10-15 m with a JUGS ball launcher.
  Arms: Soccer Heading (Oblique)

SUMMARY:
There is growing concern for the resulting neurological and physiological outcomes from repeated head impacts in sports that do not manifest into traditional concussion symptoms. Specifically, there is evidence of immediate physiological deficits following controlled soccer heading. This study will compare the physiological changes of adolescents completing a set of soccer headers to those randomized to a set of soccer kicks to evaluate the effect of repetitive head impacts.

DETAILED DESCRIPTION:
There is limited data relating head impact biomechanics to neurological outcomes in humans. Concussion occurs from rotational loading of the head giving rise to diffuse stresses and strains in the brain tissue leading to autonomic and physiological dysfunction. Repeated head loading is common in contact sports and an integral part of soccer. It is unknown whether the same biomechanical forces from lower severity head impacts such as typical soccer heading cause temporary physiological deficits as well. Advancement of objective physiological function assessment devices allow measurement of neurological effects in the absence of diagnosed concussion. Recent soccer heading studies have evaluated neurophysiological changes pre- and post-repetitive heading. These studies have found conflicting results for the effect on neurocognitive performance immediately following a bout of heading, but consistent changes were observed in measures of vestibular balance, ocular function, and neurochemical biomarkers.

Soccer heading biomechanics studies showed that females experienced higher severity head loading, and in equivalent sports such as soccer and basketball, females have higher concussion rates. This study will compare the physiological changes of male and female adolescents completing one of two soccer heading paradigms to those randomized to kicking to evaluate the effect of repetitive head impacts. This study will relate biomechanical measures of head loading with physiological function changes associated with repeated head impacts, and compare sex-differences in biomechanical measures and physiological changes.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ages 13 to 18.
* Actively participating on a competitive soccer team.
* At least 1 year of soccer heading experience.
* Parental/guardian permission (informed consent) and child assent.

Exclusion Criteria:

* Subject sustained a concussion or spinal injury within the past 6 months or still has active symptoms from a previous injury.
* Inability to exercise because of lower-extremity orthopedic injury or significant vestibular or visual dysfunction.
* Currently taking medications that can affect autonomic function.
* Plays exclusively the goalkeeper position and does not regularly head the ball.
* Parental/guardian permission (informed consent) not obtainable or not provided.
* Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
* Subject has fixed orthodontia on upper teeth.
* Cannot understand English.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-19 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Concussion Exam immediately post intervention | Pre-intervention to 0 hours post intervention
  A standard concussion physical exam includes smooth pursuits, horizontal and vertical saccades, horizontal and vertical gaze stability, visual motion sensitivity, convergence and divergence, and tandem walk.

SECONDARY OUTCOMES:
Head linear acceleration | During Intervention
  Linear acceleration (g) of the head will be measured during soccer heading via an instrumented mouthguard equipped with a 3-axis accelerometer.
Head angular velocity | During Intervention
  Angular velocity (radians/second) of the head will be measured during soccer heading via an instrumented mouthguard equipped with a 3-axis gyroscope.
Change in Clinical Concussion Exam at up to 72 hours post intervention | Pre-intervention to between 16 and 72 hours post intervention
  A standard concussion physical exam includes smooth pursuits, horizontal and vertical saccades, horizontal and vertical gaze stability, visual motion sensitivity, convergence and divergence, and tandem walk.

OTHER OUTCOMES:
King-Devick Test | Pre-intervention, 0 hours post and up to 72 hours post intervention
  The test assesses saccadic eye movement based on rapidly naming single-digit numbers from left to right on test cards, a laptop, or a tablet.
Pupillary Light Reflex | Pre-intervention, 0 hours post and up to 72 hours post intervention
  The dilation of the pupil in response to a visual stimulus
Visual Evoked Potential | Pre-intervention, 0 hours post and up to 72 hours post intervention
  The electrical brain activity in the entire vision system measured via surface electrodes following a reverse pattern visual stimulus.
Balance | Pre-intervention, 0 hours post and up to 72 hours post intervention
  Static balance will be assessed by the Biodex BioSway while standing on firm and foam surfaces with eyes open and closed.
Neck Strength | Pre-intervention, 0 hours post and up to 72 hours post intervention
  Maximum isometric voluntary contraction for neck flexion
Muscle Activation | Pre-intervention, 0 hours post and up to 72 hours post intervention
  Electromyography of the sternocleidomastoid and trapezius muscle activation during maximum isometric voluntary contraction and soccer kicking/heading.

CONTACTS AND LOCATIONS:
Overall Officials: Kristy B Arbogast, PhD, Principal Investigator — Children's Hospital of Philadelphia; Christina L Master, MD, Study Chair — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT04810130/ICF_000.pdf